CLINICAL TRIAL: NCT04100044
Title: A Pilot Study to Assess Adherence of an Exercise Prescription in Elderly Multiple Myeloma Patients
Brief Title: Exercise Prescription for the Improvement of Quality of Life in Elderly Patients With Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 19G.514; JT 13791 (Other: JeffTrial Number)
Record Dates: First submitted 2019-09-04; First posted 2019-09-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health Services Research (physical therapist, exercise) (Experimental): Patients meet with a physical therapist on day 0 and at 3 and 6 months and receive a personalized home exercise intervention consisting of aerobic and resistance training for 6 months. Patients also receive face-to-face sessions, video chats, or text message check-ins with physical therapist weekly for 6 weeks and then every other week for up to 24 weeks.
  Interventions: Other: Exercise Counseling; Behavioral: Exercise Intervention; Other: Questionnaire administration; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Exercise Counseling — Meet with physical therapist
Behavioral: Exercise Intervention — Receive personalized home exercise intervention
Other: Questionnaire administration — Ancillary studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This trial studies how well exercise prescription works in improving quality of life in elderly patients with multiple myeloma. Engaging and adhering to an exercise program may improve functional status and quality of life and decrease pain and skeletal-related events. This study is being done to see if elderly patients with multiple myeloma can participate in a physical activity program.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the ability for elderly multiple myeloma patients to maintain a personalized exercise regimen and activity level for a period of 6 months.

SECONDARY OBJECTIVE:

I. Assess changes in biometric data.

EXPLORATORY OBJECTIVE I. Evaluate changes in bone metabolism markers as a result of exercise.

OUTLINE:

Patients meet with a physical therapist on day 0 and at 3 and 6 months and receive a personalized home exercise intervention consisting of aerobic and resistance training for 6 months. Patients also receive face-to-face sessions, video chats, or text message check-ins with physical therapist weekly for 6 weeks and then every other week for up to 24 weeks.

After completion of study, patients are followed up every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple myeloma
* If patients are undergoing an autologous stem cell transplant, then they will be enrolled after their transplant so that there is not an interruption in the study period
* Patients are eligible whether or not they have lytic bone lesions

  * If they do have lytic lesions, the lesions must be low risk for fracture (low risk by Mirel's score or less than 50% of vertebral body height)
  * If patients are high risk for bone fracture, they must undergo bone stabilization prior to being considered for enrollment
  * Patients will have to be at least 6 weeks from date of stabilization
* Provide signed and dated informed consent form
* Willing to comply with all study procedures and be available for the duration of the study
* Subjects need to be within 24 months of their multiple myeloma diagnosis
* Subject must be able to stand and walk to perform baseline assessments
* Subjects must be able to text message (will need cell phone)
* Need to limit to able to read and understand English as video visit capability is only in English at this point in time and multiple questionnaires will not be translated into other languages

Exclusion Criteria:

* Presence of lytic lesions that cannot undergo appropriate stabilization
* Anything that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study
* Non English speaking
* Diagnosed greater than 24 months prior to screening

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-05-27 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Physical activity adherence | Up to 6 months
  Will be measured at each assessment using an Actigraph tri-axial hip-worn accelerometers, worn for 7 days at each assessment point, supplemented with patient self-report of exercise in the past 7 days using a physical activity recall to differentiate subtypes of physical activity. Will estimate the proportion of participants who maintained their target level, along with an exact 95% confidence interval. We will use an exact binomial test to assess whether adherence exceeds 50%. Adherence to the exercise prescriptions will be measured with the absolute and relative increase from baseline in min/week of aerobic and resistance exercise at 3 months and 6 months (benchmark: min/week of exercise changes by > 100% and a minimum of 90 min/week at 6 months). The percent of prescribed minutes of exercise performed at 3 and 6 months also will be calculated with goal of adherence greater than 50%.
Retention | Up to 6 months
  Will be measured by percent number of days the patient wears the provided FitBit during the 6-month period.

SECONDARY OUTCOMES:
Change in short physical performance battery protocol | Baseline up to 6 months
  The Short Physical Performance Battery Protocol is a test consisting of three sections (Balance, Gait Speed, and Chair Stand). The score for the Short Physical Performance Battery Protocol is scored as a total of the points earned in each section. Scores range from a total of 0 to 12 points.
  Will use methods for paired data to estimate the mean difference, along with a 95% confidence interval. Will carry out additional analyses to assess the change of these outcomes over time, utilizing the repeated measurements obtained at all timepoints. Will use mixed-effects regression for all analyses.
Change in 6 minute walk test | Baseline up to 6 months
  Will use methods for paired data to estimate the mean difference, along with a 95% confidence interval. Will carry out additional analyses to assess the change of these outcomes over time, utilizing the repeated measurements obtained at all timepoints. Will use mixed-effects regression for all analyses.
Change in grip strength | Baseline up to 6 months
  Grip strength will be measured using a dynamometer, which gives results in kg of force. Will use methods for paired data to estimate the mean difference, along with a 95% confidence interval. Will carry out additional analyses to assess the change of these outcomes over time, utilizing the repeated measurements obtained at all timepoints. Will use mixed-effects regression for all analyses.
Change in Mini-Balance Evaluation Systems Test | Baseline up to 6 months
  Will use methods for paired data to estimate the mean difference, along with a 95% confidence interval. Will carry out additional analyses to assess the change of these outcomes over time, utilizing the repeated measurements obtained at all timepoints. Will use mixed-effects regression for all analyses.
Change in frailty score | Baseline up to 6 months
  Will use methods for paired data to estimate the mean difference, along with a 95% confidence interval. Will carry out additional analyses to assess the change of these outcomes over time, utilizing the repeated measurements obtained at all timepoints. Will use mixed-effects regression for all analyses.

OTHER OUTCOMES:
Change in bone metabolism markers | Baseline up to 6 months
  Will include bone specific alkaline phosphatase, tartrate resistant acid phosphatase, C-terminal telopeptide fragment of type 1 collagen, and metabolomics signatures. Will trend metabolomics signatures as described above over time for individual participants and relate them to exercise adherence. Samples will be randomized in order to avoid machine drifts. All measurements will be carried out at least in triplicate and the false discovery rate will be used for hypothesis testing to determine the rate of type I errors when conducting multiple comparisons.
Change in pain level | Baseline up to 6 months
  Will be measured by Brief Pain Inventory. There are 9 total questions consisting of: 1 diagram, 1 yes/no, 1 item to list pain medications/treatments, 5 questions with an 11-point rating scale, and one question with sub-items A-G with an 11-point rating scale for each sub-item. Scored as follows: Pain Severity Score = Mean of items 3-6 (pain at its worst, pain at its least, average Pain Interference Score = Mean of items 9A-9G (interference of pain with: general activity, mood, walking, normal work, relations, sleep, enjoyment of life).
Change in quality of life (QOL) | Baseline up to 6 months
  Will be measured by European Organization of Research and Treatment of Cancer - QOL survey. There are 20 questions on a 4 point scale. Scores range from 0 to 100.
Participant satisfaction | At 6 months
  This is an 8 question survey with likert scale answers. Will be measured by a participant satisfaction questionnaire as well as open feedback questions to guide future studies.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Binder, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No